CLINICAL TRIAL: NCT00850447
Title: Cognitive Remediation in PTSD
Brief Title: Cognitive Remediation in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: VISN 3 Mental Illness Research, Education and Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rachel Yehuda, PhD, Professor of Neuroscience and Psychiatry, Bronx VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALT-08-045
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic stress disorder; Cognition; Neuropsychological Tests
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Remediation Therapy (Experimental)
  Interventions: Other: Cognitive Remediation Therapy
- Videogames (Placebo Comparator)
  Interventions: Other: Videogame

INTERVENTIONS:
Other: Cognitive Remediation Therapy — Cognitive Remediation Therapy (CRT) is a standardized intervention that involves performing cognitive exercises to improve attention, processing speed, and memory through practice. Participants will have one 60-minute CRT session each week for ten weeks. The CRT to be used in the proposed study is CogPack (version 6.0 Marker Software, Mannheim Germany). CogPack demonstrates flexibility in terms of developing a targeted intervention plan based on the levels of baseline cognitive impairment. There are approximately 6 different exercises presented in each training session, with the starting level of difficulty individualized on the basis of baseline neuropsychological performance.
  Arms: Cognitive Remediation Therapy
Other: Videogame — Participants will play the videogame Tetris once each week for 30 minutes. Tetris is a video puzzle game that involves manipulating falling shapes. The object of the game is to manipulate these shapes, by moving them sideways or rotating them, to create a horizontal line of blocks without gaps. As the game progresses, the shapes fall faster.
  Arms: Videogames

SUMMARY:
The purpose of this study is to gather feasibility data on cognitive remediation therapy (CRT) as an alternative intervention for PTSD. CRT is a standardized intervention that involves performing cognitive exercises to improve attention, processing speed, and memory through practice. Although the primary objective will be to determine the effect of CRT on cognitive functioning in PTSD, data on PTSD symptom severity and other clinical measures will also be examined to assess whether and to what degree cognitive alterations and symptom severity might be linked. CogPack, a computer-based form of CRT, would be employed for this project. Participants will be randomized to receive CRT or to play the video game Tetris as a control condition.

DETAILED DESCRIPTION:
The effects of CRT will be examined in 30 combat veterans with current PTSD, to be randomized to either CRT or to a non-therapeutic video game. PTSD status and other clinical data will be collected via interview to include the Clinician Administered PTSD Scale; the Hamilton Depression Rating Scale; and the Structured Clinical Interview for DSM-IV (SCID). Subjects will also complete self-report measures, including the Posttraumatic Stress Disorder Checklist-Stressor Specific Version; Deployment Risk and Resilience Inventory; Combat Exposure Scale; Trauma History Questionnaire; Childhood Trauma Questionnaire; State-Trait Anxiety Inventory-State; Beck Depression Inventory-II; Post-Traumatic Cognitions Inventory; Connor-Davidson Resilience Scale; and the Inventory of Daily Living. Baseline cognitive functioning will be assessed using the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery; the vocabulary and block design tasks of the Wechsler Adult Intelligence Scale-III; the Wide Range Achievement Test-III; and the Logical Memory Test, the Letter-Number Sequencing task, and the Digit Span tasks from the Wechsler Memory Scale-III.

After evaluation, 15 subjects will be randomized to receive 10 weekly 60-minute sessions of CRT using CogPack Professional (version 8.2, Marker Software, Mannheim, Germany). Approximately six different exercises will be presented in each training session, with the starting level of difficulty individualized on the basis of baseline neuropsychological performance and difficulty level adjusted based on the subject's performance on CogPack exercises.

Another 15 subjects will be randomized to use a non-therapeutic video game, Tetris. Tetris is a video puzzle game that involves manipulating falling shapes. The object of the game is to manipulate these shapes, by moving them sideways or rotating them, to create a horizontal line of blocks without gaps. As the game progresses, the shapes fall faster. This game primarily involves using visuospatial and motor abilities, rather than memory and attentional abilities, and thus will serve as an adequate control condition to Cogpack. Subjects will use Tetris in 10 weekly 30-minute sessions.

Subjects will again complete neuropsychological and psychiatric evaluations (with the exception of the SCID) in addition to self-report measures after 10 weeks of CRT or video games. Changes from baseline will be examined in the cognitive measures as well as in PTSD symptom severity, other clinical measures, and overall functioning.

ELIGIBILITY:
Inclusion Criteria:

* Male and female combat veterans with a current diagnosis of PTSD with a minimum duration of six months
* Age 18 years and older
* Capable of understanding, reading, and writing in English

Exclusion Criteria:

* Incapable and/or unwilling to provide written informed consent prior to participation
* Less than 11 years of formal education
* The veteran, the veteran's physician, or the study physician thinks that the veteran's clinical state necessitates hospitalization
* Response of 3 or 4 on the suicidality items of the Hamilton Depression Rating Scale or an assessed serious suicide risk
* Current substance and/or alcohol abuse and/or dependence, or abuse/dependence within the previous 6 months which contraindicates participation in the judgment of the evaluating clinician
* A lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, organic mental disorder, or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning, assessed by Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery and portions of Wechsler Adult Intelligence Scale III (WAIS-III) and Wechsler Memory Scale III (WMS-III) | 10 weeks

SECONDARY OUTCOMES:
PTSD symptom severity, assessed by Clinician Administered PTSD Scale (CAPS) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Altman, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States